CLINICAL TRIAL: NCT07042386
Title: CROWN: Implementation of a Beauty Salon-Based Strategy for Blood Pressure Management Among Women
Brief Title: Implementation of a Beauty Salon-Based Strategy for Blood Pressure Management Among Women
Acronym: CROWN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00497859; 25ISA1453143 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hypertension
Keywords: Hypertension; Implementation Science; Beauty Salon; Women; Community Based Intervention; Cardiovascular Disease Prevention
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors and data analysts will be masked to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CROWN Intervention Arm (Experimental): Participants will receive in-salon blood pressure screenings by trained stylists, a home blood pressure monitor connected to a telemonitoring app, community health worker coaching, pharmacist medication support, and digital social needs screening with referrals.
  Interventions: Behavioral: CROWN Intervention
- Enhanced Usual Care Arm (Active Comparator): Participants will receive in-salon blood pressure screenings, a free Omron home monitor, printed cardiovascular health materials, and standard referrals to social and health services, without telemonitoring, coaching, or pharmacist support.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: CROWN Intervention — CROWN Intervention includes:
  1. Private BP screenings in salon "Heart Health Stations" by trained Heart Health Stylists
  2. Free Omron home BP monitor paired with a mobile app for twice-daily telemonitoring
  3. In-depth coaching sessions + monthly check-ins with a community health worker
  4. Bi-weekly medication review and adherence support by a clinical pharmacist
  5. Digital social-needs screening (AHC HRSN) with referral to community resources
  Arms: CROWN Intervention Arm
Behavioral: Enhanced Usual Care — Enhanced Usual Care include:
  1. Private BP screenings in salon "Heart Health Stations" by Heart Health Stylists
  2. Printed cardiovascular health brochures
  3. Free home blood pressure monitor (no app integration)
  4. Standard referrals to social and health services
  Arms: Enhanced Usual Care Arm

SUMMARY:
CROWN is a two-arm, cluster-randomized pilot trial testing the feasibility and preliminary efficacy of a salon-based cardiovascular intervention - training stylists as Heart Health Stylists to conduct in-salon blood pressure screenings, home monitoring with telehealth support, community health-worker coaching, and pharmacist-led medication management - among Black and Hispanic women with hypertension.

DETAILED DESCRIPTION:
CROWN is a six-month, cluster-randomized pilot trial enrolling approximately 12 beauty salons. In intervention salons, trained Heart Health Stylists provide weekly private blood pressure screenings. Participants recruited from the intervention salons will receive a home blood pressure monitor linked to a mobile app, as well as community health worker coaching sessions and pharmacist medication support. Participants in the enhanced usual care salons will receive only printed educational materials and a home blood pressure monitor. Eligibility (age ≥18, self-identified Black or Hispanic, Systolic Blood Pressure (SBP) ≥130/80) will be confirmed via three standardized BP measurements, medical history review, and medication assessment in private salon alcoves or by phone. Assessments at baseline, 12, and 24 weeks include seated blood pressure (BP), weight, point-of-care hemoglobin A1c, and lipid panels, as well as surveys of health behaviors and social needs. Participants will receive gift cards, and retain the home monitor at the end of the study. The primary outcome is the change in systolic blood pressure; secondary outcomes include blood pressure control rates, adherence, lifestyle behaviors, and social needs resolution, with end-of-study qualitative interviews assessing acceptability.

ELIGIBILITY:
Inclusion Criteria:

Women are eligible if:

* At least 18 years old
* Self-identify as Black/African American or Hispanic
* Have an average seated systolic blood pressure of 130 mmHg or higher on initial salon screening, and
* Have visited the participating salons at least twice in the past six months.

Exclusion Criteria:

Women are excluded if:

* Pregnant or planning pregnancy during the study period
* Have end-stage renal disease requiring dialysis
* Have serious medical conditions limiting life expectancy to less than 12 months
* Currently participating in other cardiovascular intervention studies
* Have severe cognitive impairment, impeding informed consent
* Unable to operate blood pressure monitoring equipment after training
* Plan to relocate outside the study area within 6 months
* Have documented adverse reactions to blood pressure cuff usage.

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility is limited to individuals aged 18 years or older, who self-identify as women regardless of sex assigned at birth, and who self-identify as Black/African American or Hispanic.
Enrollment: 144 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in systolic blood pressure | Baseline, 3 months, 6 months
  Mean change in systolic blood pressure as assessed by standardized American Heart Association (AHA)-guided automated measurements in the salon and at home (average of three seated readings after 5 minutes' rest).

SECONDARY OUTCOMES:
Change in Hemoglobin A1c | Baseline, 3 months, 6 months
  Hemoglobin A1c by finger-stick point of care testing (POCT)
Change in weight, measured in pounds | Baseline, 3 months, 6 months
  Change in weight via calibrated scales
Change in lipids level | Baseline, 3 months, 6 months
  Change in lipids level by finger-stick point of care testing (POCT)
Change in Percent Body Fat | Baseline, 3 months, 6 months
  Change in percent body fat via calibrated scales
Mean change in diastolic blood pressure | Baseline, 3 months, 6 months
  Mean change in diastolic blood pressure as assessed by standardized American Heart Association (AHA)-guided automated measurements in the salon and at home (average of three seated readings after 5 minutes' rest).

OTHER OUTCOMES:
Change in Number of times health-related social resources were accessed | Baseline, 3 months, 6 months
  Social resource utilization assessed by the AHC Health-Related Social Needs (HRSN) digital screening tool
Change in Health-related quality of life | Baseline, 6 months
  Measured with the Patient-Reported Outcomes Measurement Information System (PROMIS)-29 instrument. Score ranges from 4-20, where a higher score correlates to better outcome.
Change in Patient activation | Baseline, 6 months
  Assessed via the Patient Activation Measure-13 (PAM-13). Score of 0-100 where higher scores indicate a better outcome
Change in Medication adherence | Baseline, 6 months
  Measured with the Hill-Bone Medication Adherence Scale. The total score ranges from 14 to 56. 14 is the worse adherence and 56 is the best adherence.
Change in Self-efficacy | Baseline, 6 months
  Assessed using the New Self-Efficacy Scale (Score Range: 1-5; Higher scores are better)
Implementation fidelity | 6 months
  Implementation fidelity will be evaluated through adherence to intervention protocols. Reporting the number of salons that completed the study.
Implementation fidelity | 6 months
  Implementation fidelity will be evaluated through adherence to intervention protocols. Reporting the number of deviations per salon.
Adoption | 6 months
  Adoption will be measured by the proportion of invited salons and stylists who engage with the intervention.
Program Cost effectiveness | 6 months
  Program costs, including expenses for stylist training, salon support, Community Health Worker (CHW) time, and technology infrastructure, will be tracked. Incremental Cost-Effectivness Ratio be reported. The ratio is the additional cost of one intervention compared to another, divided by the difference in their health outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Oluwabunmi Ogungbe, PhD, MPH, RN, Principal Investigator — Johns Hopkins School of Nursing
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States